CLINICAL TRIAL: NCT00465816
Title: Non-inferiority of GSK Biologicals' Meningococcal Vaccine 134612 Given Concomitantly With GSK Biologicals' Twinrix™ Versus 134612 Alone and Twinrix™ Alone in Healthy Subjects Aged 11 Through 17 Years.
Brief Title: Primary Study to Demonstrate Non-inferiority and Immunogenicity of GSK Biologicals' Meningococcal Vaccine 134612
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 109063
Record Dates: First submitted 2007-04-24; First posted 2007-04-25 (Estimated); Results first posted 2012-05-22 (Estimated); Last update posted 2018-06-08 (Actual); Status verified 2016-11

CONDITIONS: Infections, Meningococcal
Keywords: non-inferiority; adolescents; meningococcal vaccine
MeSH Terms: conditions — Meningococcal Infections | interventions — twinrix

ARMS (3):
- Nimenrix + Twinrix Group (Experimental): Subjects received 1 dose of Nimenrix™ vaccine at Month 0 and 1 dose of Twinrix™ vaccine at Months 0, 1 and 6.
  Interventions: Biological: Nimenrix (Meningococcal vaccine 134612); Biological: Twinrix
- Nimenrix Group (Active Comparator): Subjects received 1 dose of Nimenrix™ vaccine at Month 0.
  Interventions: Biological: Nimenrix (Meningococcal vaccine 134612)
- Twinrix Group (Active Comparator): Subjects received 1 dose of Twinrix™ vaccine at Months 0, 1 and 6.
  Interventions: Biological: Twinrix

INTERVENTIONS:
Biological: Nimenrix (Meningococcal vaccine 134612) — Single dose intramuscular injection
  Arms: Nimenrix + Twinrix Group; Nimenrix Group
Biological: Twinrix — 3-dose intramuscular injection. Twinrix Adult will be administered to subjects aged 16 years and above and Twinrix Junior will be administered to subjects aged from 11 years up to and including 15 years of age.
  Arms: Nimenrix + Twinrix Group; Twinrix Group

SUMMARY:
This study will demonstrate the non-inferiority of GSK Biologicals' meningococcal vaccine 134612 when given in an experimental co-administration versus vaccine 134612 alone and versus the experimental co-administration alone in healthy subjects aged 11 through 17 years. There will be 3 groups in this study.

DETAILED DESCRIPTION:
All subjects of groups A and B will have 4 blood samples taken, all subjects of group C will have 3 blood samples taken.

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, September 2007.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that they and/or their parents/guardians can and will comply with the requirements of the protocol
* A male or female between, and including, 11 and 17 years of age at the time of the first dose of vaccine.
* Written informed consent obtained from the subject/ from the parent or guardian of the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Previously completed routine childhood vaccinations to the best of his/her/the parents'/guardians' knowledge.
* If the subject is female and of childbearing potential, she must practice adequate contraception for 30 days prior to vaccination, have a negative pregnancy test and continue such precautions for two months after completion of the vaccination series.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Planned administration/ administration of a vaccine not foreseen by the study protocol within one month of the dose of vaccine.
* Previous vaccination with meningococcal polysaccharide vaccine of serogroup A, C, W-135 and/or Y within the last five years.
* Previous vaccination with meningococcal polysaccharide conjugate vaccine of serogroup A, C, W-135 and/or Y.
* Previous vaccination with tetanus toxoid within the last month.
* Previous vaccination with hepatitis A and/or hepatitis B vaccine.
* Seropositivity for hepatitis A IgG, hepatitis B surface antigen, hepatitis B core antibody and/or hepatitis B surface antigen at screening.
* History of hepatitis A, hepatitis B and/or Neisseria meningitidis infection.
* Known exposure to hepatitis A and/or hepatitis B virus within three months preceding the first dose of study vaccine.
* Any confirmed or suspected immunosuppressive or immunodeficient condition (congenital or secondary), including human immunodeficiency virus (HIV) infection, based on medical history and physical examination.
* A family history of congenital or hereditary immunodeficiency, until the immune competence of the potential vaccine recipient is demonstrated.
* History of reactions or allergic disease likely to be exacerbated by any component of either vaccine.
* Major congenital defects or serious chronic illness.
* Acute disease at the time of enrolment.
* Administration of immunoglobulins and/or any blood products within the three months preceding the dose of study vaccine or planned administration during the study period.
* Pregnant or lactating female.
* History of chronic alcohol consumption and/or drug abuse.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 611 (Actual)
Dates: Start 2007-04-11; Primary Completion 2008-04-28 (Actual); Study Completion 2008-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (6):
- GSK Investigational Site, Aarhus N, Denmark
- Sweden (5):
  - GSK Investigational Site, Karlskrona
  - GSK Investigational Site, Linköping
  - GSK Investigational Site, Malmo
  - GSK Investigational Site, Örebro
  - GSK Investigational Site, Umeå

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Ostergaard L, Silfverdal SA, Berglund J, Flodmark CE, West C, Bianco V, Baine Y, Miller JM. A tetravalent meningococcal serogroups A, C, W-135, and Y tetanus toxoid conjugate vaccine is immunogenic and well-tolerated when co-administered with Twinrix((R)) in subjects aged 11-17 years: an open, randomised, controlled trial. Vaccine. 2012 Jan 17;30(4):774-83. doi: 10.1016/j.vaccine.2011.11.051. Epub 2011 Nov 19. PMID 22107850
- [Background] Ostergaard L et al. The Candidate meningococcal serogroups A, C, W-135, Y tetanus toxoid conjugated vaccine (MenACWY-TT) co-administered with a combined hepatitis A and B vaccine (HepA/B) is immunogenic with an acceptable safety profile in subjects aged 11-17 Years. Abstract presented at the 3rd Northern European Conference on Travel Medicine (NECTM). Hamburg, Germany, 26-29 May 2010.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Dataset Specification: 109063 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 109063 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 109063 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 109063 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 109063 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 109063 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 109063 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: During the screening the following was performed: informed consent was obtained and signed from parents or guardians of subjects, check for inclusion/exclusion criteria and contraindications/precautions was performed, and medical history of subjects was collected.
Groups:
- Nimenrix + Twinrix Group: Subjects received 1 dose of Nimenrix vaccine at Month 0 and 1 dose of Twinrix vaccine at Months 0, 1 and 6.
- Nimenrix Group: Subjects received 1 dose of Nimenrix vaccine at Month 0.
- Twinrix Group: Subjects received 1 dose of Twinrix vaccine at Months 0, 1 and 6.
Period: Overall Study
Arm/Group | Nimenrix + Twinrix Group | Nimenrix Group | Twinrix Group
Started | 367 | 122 | 122
Completed | 367 | 122 | 120
Not Completed | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nimenrix + Twinrix Group | Nimenrix Group | Twinrix Group | Total
Number analyzed (Participants) | 367 | 122 | 122 | 611
Age, Continuous [Mean (Standard Deviation); unit: Years] | 14.3 (1.89) | 14.3 (1.84) | 14.3 (1.94) | 14.3 (1.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 195 | 61 | 68 | 324
  Male | 172 | 61 | 54 | 287
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African heritage/African American | 1 | 0 | 0 | 1
  Asian - central/south Asian heritage | 1 | 2 | 0 | 3
  Asian - east Asian heritage | 2 | 2 | 0 | 4
  Asian - south east Asian heritage | 0 | 0 | 1 | 1
  White - Arabic/north African heritage | 1 | 1 | 0 | 2
  White - Caucasian/European heritage | 361 | 117 | 121 | 599
  Not specified | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Meningococcal Polysaccharide A Serum Bactericidal Antibodies/Assay, Using Baby Rabbit Complement for Assay (rSBA-MenA), rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Titers
Description: The rSBA titers were expressed as geometric mean titers (GMTs).
Time Frame: At 1 month after vaccination with Nimenrix vaccine (Month 1)
Population: The analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity post Dose 1 including all evaluable subjects for whom immunogenicity data were available for the considered time point(s), only on those groups of subjects that received the Nimenrix vaccine.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Nimenrix + Twinrix Group | Nimenrix Group
Number analyzed (Participants) | 360 | 115
Titer
  rSBA-MenA: number analyzed (Participants) | 353 | 113
  rSBA-MenA | 5263.9 [4818.0 to 5751.0] | 5211.7 [4509.8 to 6022.8]
  rSBA-MenC | 4344.6 [3800.3 to 4966.8] | 4926.9 [3684.8 to 6587.7]
  rSBA-MenW-135 | 8922.1 [8278.4 to 9615.9] | 8987.7 [7628.9 to 10588.6]
  rSBA-MenY | 9291.5 [8537.7 to 10111.9] | 9492.8 [8172.4 to 11026.6]
Statistical Analysis 1: Comparison: Nimenrix + Twinrix Group vs Nimenrix Group; To assess the Non-inferiority in term of rSBA-MenA GMT of the Nimenrix + Twinrix group compared to Nimenrix one, two-sided 95% confidence interval (CI) from ANCOVA model on the GMTs ratio (Nimenrix+Twinrix group over Nimenrix group) was computed. The model was adjusted for age strata and baseline titre; Test type: Non-Inferiority — The lower limit of the two-sided 95% CI on the ratio of rSBA-MenA GMTs between Nimenrix + Twinrix group and (over) Nimenrix group was ≥ 0.5; ANCOVA; Adjusted GMT ratio = 0.99, 95% CI 2-sided [0.8 to 1.22]
Statistical Analysis 2: Comparison: Nimenrix + Twinrix Group vs Nimenrix Group; To assess the Non-inferiority in term of rSBA-MenC GMT of the Nimenrix+Twinrix group compared to Nimenrix one, Two-sided 95% CI from ANCOVA model on the GMTs ratio (Nimenrix+Twinrix group over Nimenrix group) was computed. The model was adjusted for age strata and baseline titre; Test type: Non-Inferiority — The lower limit of the two-sided 95% CI on the ratio of rSBA-MenC GMTs between Nimenrix + Twinrix group and (over) Nimenrix group was ≥ 0.5; ANCOVA; Adjusted GMT ratio = 0.91, 95% CI 2-sided [0.68 to 1.21]
Statistical Analysis 3: Comparison: Nimenrix + Twinrix Group vs Nimenrix Group; To assess the Non-inferiority in term of rSBA-MenW-135 GMT of the Nimenrix+Twinrixg roup compared to Nimenrix one, Two-sided 95% CI from ANCOVA model on the GMTs ratio (Nimenrix+Twinrix group over Nimenrix group) was computed. The model was adjusted for age strata and baseline titre; Test type: Non-Inferiority — The lower limit of the two-sided 95% CI on the ratio of rSBA-MenW-135 GMTs between Nimenrix + Twinrix group and (over) Nimenrix group was ≥ 0.5; ANCOVA; Adjusted GMT ratio = 1.02, 95% CI 2-sided [0.87 to 1.19]
Statistical Analysis 4: Comparison: Nimenrix + Twinrix Group vs Nimenrix Group; To assess the Non-inferiority in term of rSBA-MenY GMT of the Nimenrix+Twinrix group compared to Nimenrix one, Two-sided 95% CI from ANCOVA model on the GMTs ratio (Nimenrix+Twinrix group over Nimenrix group) was computed. The model was adjusted for age strata and baseline titre; Test type: Non-Inferiority — The lower limit of the two-sided 95% CI on the ratio of rSBA-MenY GMTs between Nimenrix + Twinrix group and (over) Nimenrix group was ≥ 0.5; ANCOVA; Adjusted GMT ratio = 1.01, 95% CI 2-sided [0.85 to 1.19]

2. Primary Outcome: Number of Subjects Seroconverted for Hepatitis A
Description: A seroconverted subject was defined as a subject with anti-Hepatitis A virus (HAV) antibody concentration greater than or equal to 15 milli-International Units per Milliliter (mIU/mL) in previously seronegative subjects.
Time Frame: At 1 month after the third dose of Twinrix vaccine (Month 7)
Population: The analysis was performed on the According-to-Protocol cohort for immunogenicity post Dose 2 and 3 including all evaluable subjects for whom immunogenicity data were available for the considered time point(s), only on initially seronegative subjects in those groups that received the Twinrix vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Twinrix Group | Twinrix Group
Number analyzed (Participants) | 321 | 95
Participants | 321 | 95
Statistical Analysis 1: Comparison: Nimenrix + Twinrix Group vs Twinrix Group; To assess the Non-inferiority of the Nimenrix+Twinrix group compared to Twinrix one, two-sided standardized asymptotic 95% CI for the difference in seroconversion rates for hepatitis A (Nimenrix+Twinrix group minus Twinrix group) was computed; Test type: Non-Inferiority — The lower limit of the two-sided standardised asymptotic 95% CI for group difference (Nimenrix+Twinrix group minus Twinrix group) in the percentage of subjects with vaccine seroconversion was ≥ pre-defined clinical limit of -10%; Percentage difference = 0, 95% CI 2-sided [-1.19 to 3.9]

3. Primary Outcome: Number of Subjects Seroprotected for Hepatitis B
Description: A seroprotected subject was defined as a subject with anti-Hepatitis B surface antigen (HBs) antibody concentration greater than or equal to 10 milli-International Units per Milliliter (mIU/mL).
Time Frame: At 1 month after the third dose of Twinrix vaccine (Month 7)
Population: The analysis was performed on the According-to-Protocol cohort for immunogenicity post Dose 2 and 3 including all evaluable subjects for whom immunogenicity data were available for the considered time point(s), only on those groups of subjects that received the Twinrix vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Twinrix Group | Twinrix Group
Number analyzed (Participants) | 330 | 97
Participants | 327 | 97
Statistical Analysis 1: Comparison: Nimenrix + Twinrix Group vs Twinrix Group; To assess the Non-inferiority of the Nimenrix+Twinrix group compared to the Twinrix one, two-sided standardized asymptotic 95% CI for the difference in seroprotection rates for hepatitis B (Nimenrix+Twinrix group minus Twinrix group) was computed; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Percentage difference = -0.91, 95% CI 2-sided [-2.64 to 2.92]

4. Secondary Outcome: Number of Subjects With a Vaccine Response to MenA, MenC, MenY and MenW-135
Description: Vaccine response is defined as an rSBA titer of at least 1:32 in subjects initially seronegative [rSBA titer below1:8] and as a 4-fold increase in titer in subjects initially seropositive [rSBA titre greater than or equal to 1:8].
Time Frame: At 1 month after vaccination with Nimenrix vaccine (Month 1)
Population: The analysis was performed on the According-to-Protocol cohort for immunogenicity post Dose 1 including all evaluable subjects for whom immunogenicity data were available for the considered time point(s), only on those groups of subjects that received the Nimenrix vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Twinrix Group | Nimenrix Group
Number analyzed (Participants) | 355 | 114
Participants
  rSBA-MenA: number analyzed (Participants) | 261 | 84
  rSBA-MenA | 246 | 76
  rSBA-MenC: number analyzed (Participants) | 355 | 112
  rSBA-MenC | 333 | 101
  rSBA-MenW-135: number analyzed (Participants) | 349 | 114
  rSBA-MenW-135 | 346 | 112
  rSBA-MenY: number analyzed (Participants) | 354 | 113
  rSBA-MenY | 335 | 105

5. Secondary Outcome: Number of Subjects With rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Titers Above Predefined Cut-off Values
Description: The cut-off values assessed were greater than or equal to (≥) 1:8 and ≥ 1:128.
Time Frame: Prior to and 1 month after vaccination with Nimenrix vaccine (Months 0 and 1)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Twinrix Group | Nimenrix Group
Number analyzed (Participants) | 360 | 115
Participants
  rSBA-MenA ≥ 1:8 [Month 0]: number analyzed (Participants) | 266 | 85
  rSBA-MenA ≥ 1:8 [Month 0] | 105 | 33
  rSBA-MenA ≥ 1:8 [Month 1]: number analyzed (Participants) | 353 | 113
  rSBA-MenA ≥ 1:8 [Month 1] | 352 | 113
  rSBA-MenC ≥ 1:8 [Month 0]: number analyzed (Participants) | 355 | 112
  rSBA-MenC ≥ 1:8 [Month 0] | 187 | 67
  rSBA-MenC ≥ 1:8 [Month 1] | 359 | 114
  rSBA-MenW-135 ≥ 1:8 [Month 0]: number analyzed (Participants) | 349 | 114
  rSBA-MenW-135 ≥ 1:8 [Month 0] | 277 | 96
  rSBA-MenW-135 ≥ 1:8 [Month 1] | 360 | 115
  rSBA-MenY ≥ 1:8 [Month 0]: number analyzed (Participants) | 354 | 113
  rSBA-MenY ≥ 1:8 [Month 0] | 275 | 95
  rSBA-MenY ≥ 1:8 [Month 1] | 359 | 115
  rSBA-MenA ≥ 1:128 [Month 0]: number analyzed (Participants) | 266 | 85
  rSBA-MenA ≥ 1:128 [Month 0] | 91 | 30
  rSBA-MenA ≥ 1:128 [Month 1]: number analyzed (Participants) | 353 | 113
  rSBA-MenA ≥ 1:128 [Month 1] | 352 | 113
  rSBA-MenC ≥ 1:128 [Month 0]: number analyzed (Participants) | 355 | 112
  rSBA-MenC ≥ 1:128 [Month 0] | 122 | 44
  rSBA-MenC ≥ 1:128 [Month 1] | 358 | 113
  rSBA-MenW-135 ≥ 1:128 [Month 0]: number analyzed (Participants) | 349 | 114
  rSBA-MenW-135 ≥ 1:128 [Month 0] | 180 | 64
  rSBA-MenW-135 ≥ 1:128 [Month 1] | 359 | 115
  rSBA-MenY ≥ 1:128 [Month 0]: number analyzed (Participants) | 354 | 113
  rSBA-MenY ≥ 1:128 [Month 0] | 218 | 80
  rSBA-MenY ≥ 1:128 [Month 1] | 359 | 115

6. Secondary Outcome: Anti-PSA (Polysaccharide A), Anti-PSC (Polysaccharide C), Anti-PSW-135 (Polysaccharide W-135), and Anti-PSY (Polysaccharide Y) Antibody Concentrations
Description: Concentrations were provided as Geometric Mean Concentrations expressed as micrograms per milliliter (µg/mL).
Time Frame: Prior to and 1 month after vaccination with Nimenrix vaccine (Months 0 and 1)
Population: The analysis was performed on the ATP cohort for immunogenicity post Dose 1, only on those groups of subjects that received Nimenrix. A randomized subset of half of the subjects had sera tested by Enzyme-linked Immunosorbent assay (ELISA) for anti-PSA and anti-PSC antibodies while the other half were tested for anti PSW-135 and anti-PSY antibodies.
Measure: Geometric Mean (95% Confidence Interval); unit: micrograms per milliliter (µg/mL)
Arm/Group | Nimenrix + Twinrix Group | Nimenrix Group
Number analyzed (Participants) | 180 | 58
micrograms per milliliter (µg/mL)
  Anti-PSA [Month 0]: number analyzed (Participants) | 176 | 55
  Anti-PSA [Month 0] | 0.25 [0.21 to 0.30] | 0.24 [0.19 to 0.31]
  Anti-PSA [Month 1]: number analyzed (Participants) | 179 | 56
  Anti-PSA [Month 1] | 27.23 [22.91 to 32.38] | 18.47 [12.02 to 28.38]
  Anti-PSC [Month 0]: number analyzed (Participants) | 176 | 55
  Anti-PSC [Month 0] | 0.22 [0.19 to 0.26] | 0.26 [0.19 to 0.35]
  Anti-PSC [Month 1]: number analyzed (Participants) | 180 | 55
  Anti-PSC [Month 1] | 18.58 [15.44 to 22.37] | 21.15 [14.87 to 30.09]
  Anti-PSW-135 [Month 0]: number analyzed (Participants) | 176 | 58
  Anti-PSW-135 [Month 0] | 0.19 [0.17 to 0.21] | 0.16 [0.15 to 0.17]
  Anti-PSW-135 [Month 1]: number analyzed (Participants) | 178 | 58
  Anti-PSW-135 [Month 1] | 6.78 [5.52 to 8.32] | 6.72 [4.62 to 9.76]
  Anti-PSY [Month 0]: number analyzed (Participants) | 175 | 58
  Anti-PSY [Month 0] | 0.22 [0.18 to 0.25] | 0.17 [0.14 to 0.21]
  Anti-PSY [Month 1]: number analyzed (Participants) | 180 | 55
  Anti-PSY [Month 1] | 14.04 [11.52 to 17.10] | 12.50 [8.49 to 18.41]

7. Secondary Outcome: Number of Subjects With Anti-PSA, Anti-PSC, Anti-PSW-135, and Anti-PSY Antibody Concentrations Above Pre-defined Cut-off Values
Description: The cut-off values assessed include greater than or equal to (≥) 0.3 micrograms per milliliter (µg/mL) and ≥ 2.0 µg/mL.
Time Frame: Prior to and 1 month after vaccination with Nimenrix vaccine (Months 0 and 1)
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Twinrix Group | Nimenrix Group
Number analyzed (Participants) | 180 | 58
Participants
  Anti-PSA ≥ 0.3 µg/mL [Month 0]: number analyzed (Participants) | 176 | 55
  Anti-PSA ≥ 0.3 µg/mL [Month 0] | 45 | 13
  Anti-PSA ≥ 0.3 µg/mL [Month 1]: number analyzed (Participants) | 179 | 56
  Anti-PSA ≥ 0.3 µg/mL [Month 1] | 179 | 54
  Anti-PSC ≥ 0.3 µg/mL [Month 0]: number analyzed (Participants) | 176 | 55
  Anti-PSC ≥ 0.3 µg/mL [Month 0] | 32 | 13
  Anti-PSC ≥ 0.3 µg/mL [Month 1]: number analyzed (Participants) | 180 | 55
  Anti-PSC ≥ 0.3 µg/mL [Month 1] | 179 | 54
  Anti-PSW-135 ≥ 0.3 µg/mL [Month 0]: number analyzed (Participants) | 176 | 58
  Anti-PSW-135 ≥ 0.3 µg/mL [Month 0] | 19 | 2
  Anti-PSW-135 ≥ 0.3 µg/mL [Month 1]: number analyzed (Participants) | 178 | 58
  Anti-PSW-135 ≥ 0.3 µg/mL [Month 1] | 176 | 56
  Anti-PSY ≥ 0.3 µg/mL [Month 0]: number analyzed (Participants) | 175 | 58
  Anti-PSY ≥ 0.3 µg/mL [Month 0] | 24 | 2
  Anti-PSY ≥ 0.3 µg/mL [Month 1]: number analyzed (Participants) | 180 | 55
  Anti-PSY ≥ 0.3 µg/mL [Month 1] | 178 | 54
  Anti-PSA ≥ 2.0 µg/mL [Month 0]: number analyzed (Participants) | 176 | 55
  Anti-PSA ≥ 2.0 µg/mL [Month 0] | 14 | 3
  Anti-PSA ≥ 2.0 µg/mL [Month 1]: number analyzed (Participants) | 179 | 56
  Anti-PSA ≥ 2.0 µg/mL [Month 1] | 178 | 52
  Anti-PSC ≥ 2.0 µg/mL [Month 0]: number analyzed (Participants) | 176 | 55
  Anti-PSC ≥ 2.0 µg/mL [Month 0] | 10 | 6
  Anti-PSC ≥ 2.0 µg/mL [Month 1]: number analyzed (Participants) | 180 | 55
  Anti-PSC ≥ 2.0 µg/mL [Month 1] | 176 | 53
  Anti-PSW-135 ≥ 2.0 µg/mL [Month 0]: number analyzed (Participants) | 176 | 58
  Anti-PSW-135 ≥ 2.0 µg/mL [Month 0] | 3 | 0
  Anti-PSW-135 ≥ 2.0 µg/mL [Month 1]: number analyzed (Participants) | 178 | 58
  Anti-PSW-135 ≥ 2.0 µg/mL [Month 1] | 146 | 48
  Anti-PSY ≥ 2.0 µg/mL [Month 0]: number analyzed (Participants) | 175 | 58
  Anti-PSY ≥ 2.0 µg/mL [Month 0] | 10 | 2
  Anti-PSY ≥ 2.0 µg/mL [Month 1]: number analyzed (Participants) | 180 | 55
  Anti-PSY ≥ 2.0 µg/mL [Month 1] | 172 | 51

8. Secondary Outcome: Anti-Tetanus Toxoid (TT) Antibody Concentrations
Description: Concentrations were provided as Geometric Mean Concentrations expressed as International Units per milliliter (IU/mL).
Time Frame: Prior to and 1 month after vaccination with Nimenrix vaccine (Months 0 and 1)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: International Units per milliliter
Arm/Group | Nimenrix + Twinrix Group | Nimenrix Group
Number analyzed (Participants) | 355 | 114
International Units per milliliter
  Month 0: number analyzed (Participants) | 312 | 114
  Month 0 | 0.800 [0.692 to 0.926] | 1.020 [0.795 to 1.308]
  Month 1: number analyzed (Participants) | 355 | 112
  Month 1 | 16.794 [15.318 to 18.411] | 17.252 [14.603 to 20.381]

9. Secondary Outcome: Number of Subjects With Anti-tetanus Toxoid Antibody Concentrations Above the Pre-defines Cut-off Value
Description: The cut-off value assessed was greater than or equal to 0.1 International Units per milliliter (IU/mL).
Time Frame: Prior to and 1 month after vaccination with Nimenrix vaccine (Months 0 and 1)
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Twinrix Group | Nimenrix Group
Number analyzed (Participants) | 355 | 114
Participants
  Month 0: number analyzed (Participants) | 312 | 114
  Month 0 | 293 | 111
  Month 1: number analyzed (Participants) | 355 | 112
  Month 1 | 354 | 112

10. Secondary Outcome: rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Titers at Month 7
Description: The rSBA titers were expressed as geometric mean titers.
Time Frame: At 7 months after vaccination with Nimenrix (At Month 7)
Population: The analysis was performed on the According-to-Protocol cohort for immunogenicity post Dose 2 and 3 including all evaluable subjects for whom immunogenicity data were available for the considered time point(s), only on those groups of subjects that received the Nimenrix vaccine.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Nimenrix + Twinrix Group | Nimenrix Group
Number analyzed (Participants) | 334 | 112
Titer
  rSBA-MenA: number analyzed (Participants) | 332 | 108
  rSBA-MenA | 2121.6 [1913.5 to 2352.2] | 2298.3 [1909.0 to 2767.0]
  rSBA-MenC | 952.4 [826.2 to 1097.8] | 1053.9 [803.1 to 1382.9]
  rSBA-MenW-135 | 3283.4 [2998.4 to 3595.4] | 3497.7 [3008.0 to 4067.2]
  rSBA-MenY | 4432.7 [4027.4 to 4878.8] | 4455.6 [3821.4 to 5195.1]

11. Secondary Outcome: Number of Subjects With rSBA-MenA, rSBA-MenC, rSBA-MenW-135 and rSBA-MenY Titers Above Predefined Cut-off Values at Month 7
Description: The cut-off values assessed were greater than or equal to (≥) 1:8 and ≥ 1:128.
Time Frame: At 7 months after vaccination with Nimenrix (At Month 7)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Twinrix Group | Nimenrix Group
Number analyzed (Participants) | 334 | 112
Participants
  rSBA-MenA ≥ 1:8: number analyzed (Participants) | 332 | 108
  rSBA-MenA ≥ 1:8 | 330 | 107
  rSBA-MenC ≥ 1:8 | 332 | 110
  rSBA-MenW-135 ≥ 1:8 | 334 | 112
  rSBA-MenY ≥ 1:8 | 333 | 112
  rSBA-MenA ≥ 1:128: number analyzed (Participants) | 332 | 108
  rSBA-MenA ≥ 1:128 | 329 | 107
  rSBA-MenC ≥ 1:128 | 318 | 108
  rSBA-MenW-135 ≥ 1:128 | 333 | 112
  rSBA-MenY ≥ 1:128 | 332 | 112

12. Secondary Outcome: Anti-PSA, Anti-PSC, Anti-PSW-135 and Anti-PSY Antibody Concentrations at Month 7
Description: Concentrations were provided as Geometric Mean Concentrations expressed as micrograms per milliliter (µg/mL).
Time Frame: At 7 months after vaccination with Nimenrix (At Month 7)
Population: The analysis was performed on the ATP cohort for immunogenicity post Dose 2 and 3, only on those groups of subjects that received Nimenrix. A randomized subset of half of the subjects had sera tested by ELISA for anti-PSA and anti-PSC antibodies while the other half were tested for anti PSW-135 and anti-PSY antibodies.
Measure: Geometric Mean (95% Confidence Interval); unit: micrograms per milliliter (µg/mL)
Arm/Group | Nimenrix + Twinrix Group | Nimenrix Group
Number analyzed (Participants) | 167 | 56
micrograms per milliliter (µg/mL)
  Anti-PSA: number analyzed (Participants) | 163 | 56
  Anti-PSA | 4.14 [3.34 to 5.15] | 3.88 [2.44 to 6.16]
  Anti-PSC: number analyzed (Participants) | 164 | 56
  Anti-PSC | 3.28 [2.60 to 4.14] | 4.15 [2.59 to 6.67]
  Anti-PSW-135 | 2.46 [1.99 to 3.05] | 3.08 [2.11 to 4.50]
  Anti-PSY: number analyzed (Participants) | 161 | 54
  Anti-PSY | 3.76 [2.95 to 4.78] | 4.28 [2.90 to 6.31]

13. Secondary Outcome: Number of Subjects With Anti-PSA, Anti-PSC, Anti-PSW-135 and Anti-PSY Antibody Concentrations Above Pre-defined Cut-off Values at Month 7
Description: The cut-off values assessed include greater than or equal to (≥) 0.3 micrograms per milliliter (µg/mL) and ≥ 2.0 µg/mL.
Time Frame: At 7 months after vaccination with Nimenrix (At Month 7)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Twinrix Group | Nimenrix Group
Number analyzed (Participants) | 167 | 56
Participants
  Anti-PSA ≥ 0.3 µg/mL: number analyzed (Participants) | 163 | 56
  Anti-PSA ≥ 0.3 µg/mL | 160 | 52
  Anti-PSC ≥ 0.3 µg/mL: number analyzed (Participants) | 164 | 56
  Anti-PSC ≥ 0.3 µg/mL | 157 | 52
  Anti-PSW-135 ≥ 0.3 µg/mL | 157 | 51
  Anti-PSY ≥ 0.3 µg/mL: number analyzed (Participants) | 161 | 54
  Anti-PSY ≥ 0.3 µg/mL | 154 | 53
  Anti-PSA ≥ 2.0 µg/mL: number analyzed (Participants) | 163 | 56
  Anti-PSA ≥ 2.0 µg/mL | 110 | 34
  Anti-PSC ≥ 2.0 µg/mL: number analyzed (Participants) | 164 | 56
  Anti-PSC ≥ 2.0 µg/mL | 94 | 35
  Anti-PSW-135 ≥ 2.0 µg/mL | 93 | 41
  Anti-PSY ≥ 2.0 µg/mL: number analyzed (Participants) | 161 | 54
  Anti-PSY ≥ 2.0 µg/mL | 104 | 37

14. Secondary Outcome: Immunoglobulin G (IgG) Anti-HAV Antibody Concentrations
Description: Concentrations are given as Geomatric Mean Concentrations expressed as milli-Internatinal Units per Milliliter (mIU/mL).
Time Frame: Prior to the first dose (Month 0) and 1 month after the third dose of Twinrix vaccine (Month 7)
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: milli-Internatinal Units per Milliliter
Arm/Group | Nimenrix + Twinrix Group | Twinrix Group
Number analyzed (Participants) | 333 | 99
milli-Internatinal Units per Milliliter
  Month 0 | 7.9 [7.6 to 8.1] | 7.6 [7.4 to 7.9]
  Month 7: number analyzed (Participants) | 331 | 97
  Month 7 | 5876.7 [5362.9 to 6439.8] | 6739.0 [5757.4 to 7887.9]

15. Secondary Outcome: Number of Subjects With IgG Anti-HAV Antibody Concentrations Above the Pre-defined Cut-off Value
Description: The cut-off value assessed was greater than or equal to 15 milli-Internatinal Units per Milliliter (mIU/mL).
Time Frame: Prior to the first dose (Month 0) and 1 month after the third dose of Twinrix vaccine (Month 7)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Twinrix Group | Twinrix Group
Number analyzed (Participants) | 333 | 99
Participants
  Month 0 | 10 | 2
  Month 7: number analyzed (Participants) | 331 | 97
  Month 7 | 331 | 97

16. Secondary Outcome: IgG Anti-HBs Antibody Concentrations
Description: Concentrations are given as Geomatric Mean Concentrations expressed as milli-Internatinal Units per Milliliter (mIU/mL).
Time Frame: Prior to the first dose (Month 0) and 1 month after the third dose of Twinrix vaccine (Month 7)
Population: The analysis was performed on the According-to-Protocol cohort for immunogenicity including all evaluable subjects for whom immunogenicity data were available for the considered time point(s), only on those groups of subjects that received the Twinrix vaccine.
Measure: Geometric Mean (95% Confidence Interval); unit: milli-Internatinal Units per Milliliter
Arm/Group | Nimenrix + Twinrix Group | Twinrix Group
Number analyzed (Participants) | 333 | 100
milli-Internatinal Units per Milliliter
  Month 0 | 1.7 [1.6 to 1.7] | 1.7 [1.6 to 1.8]
  Month 7: number analyzed (Participants) | 330 | 97
  Month 7 | 6088.2 [4977.5 to 7446.7] | 7654.7 [5518.8 to 10617.3]

17. Secondary Outcome: Number of Subjects With IgG Anti-HB Antibody Concentrations Above the Pre-defined Cut-off Value
Description: The cut-off value assessed was greater than or equal to 10 milli-Internatinal Units per Milliliter (mIU/mL).
Time Frame: Prior to the first dose (Month 0) and 1 month after the third dose of Twinrix vaccine (Month 7)
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Twinrix Group | Twinrix Group
Number analyzed (Participants) | 333 | 100
Participants
  Month 0 | 1 | 0
  Month 7: number analyzed (Participants) | 330 | 97
  Month 7 | 327 | 97

18. Secondary Outcome: Number of Subjects Reporting Any Solicited Local Symptoms Post-meningococcal Vaccination
Description: Solicited local symptoms assessed include pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade.
Time Frame: During a 4-day period (Days 0-3) after Nimenrix vaccination
Population: The analysis was done on the Total Vaccinated Cohort including all subjects with study vaccine administered and with a completed symptom sheet. Only subjects from the groups receiving Nimenrix were assessed.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Twinrix Group | Nimenrix Group
Number analyzed (Participants) | 365 | 119
Participants
  Pain | 181 | 58
  Redness | 75 | 19
  Swelling | 71 | 18

19. Secondary Outcome: Number of Subjects Reporting Any Solicited Local Symptoms Post-Twinrix Vaccination
Description: as for outcome 18
Time Frame: During a 4-day period (Days 0-3) after each Twinrix vaccination, and across doses
Population: The analysis was done on the Total Vaccinated Cohort including all subjects with study vaccine administered and with a completed symptom sheet. Only subjects from the groups receiving Twinrix were assessed.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Twinrix Group | Twinrix Group
Number analyzed (Participants) | 366 | 122
Participants
  Any Pain, Dose 1: number analyzed (Participants) | 365 | 121
  Any Pain, Dose 1 | 143 | 52
  Any Redness, Dose 1: number analyzed (Participants) | 365 | 121
  Any Redness, Dose 1 | 36 | 9
  Any Swelling, Dose 1: number analyzed (Participants) | 365 | 121
  Any Swelling, Dose 1 | 18 | 4
  Any Pain, Dose 2: number analyzed (Participants) | 361 | 119
  Any Pain, Dose 2 | 99 | 34
  Any Redness, Dose 2: number analyzed (Participants) | 361 | 119
  Any Redness, Dose 2 | 27 | 6
  Any Swelling, Dose 2: number analyzed (Participants) | 361 | 119
  Any Swelling, Dose 2 | 12 | 5
  Any Pain, Dose 3: number analyzed (Participants) | 358 | 116
  Any Pain, Dose 3 | 143 | 41
  Any Redness, Dose 3: number analyzed (Participants) | 358 | 116
  Any Redness, Dose 3 | 30 | 14
  Any Swelling, Dose 3: number analyzed (Participants) | 358 | 116
  Any Swelling, Dose 3 | 29 | 15
  Any Pain, Across doses | 228 | 73
  Any Redness, Across doses | 63 | 19
  Any Swelling, Across doses | 49 | 19

20. Secondary Outcome: Number of Subjects Reporting Any Solicited General Symptoms
Description: Solicited general symptoms assessed include fatigue, fever (axillary temperature greater than or equal to 37.5 degrees Celcius), gastrointestinal symptoms and headache. Any = occurrence of the symptom regardless of intensity grade. Dose 1 = post-Nimenrix and post-Twinrix for the Nimenrix + Twinrix Group, post-Twinrix for the Twinrix Group and post-Nimenrix for the Nimenrix Group, Dose 2, 3 and Across doses = post-Twinrix for the Nimenrix + Twinrix Group and for the Twinrix Group.
Time Frame: During a 4-day period (Days 0-3) after each vaccine dose and across doses
Population: The analysis was done on the Total Vaccinated Cohort including all subjects with study vaccine administered and with a completed symptom sheet.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Twinrix Group | Nimenrix Group | Twinrix Group
Number analyzed (Participants) | 366 | 119 | 122
Participants
  Any Fatigue, Dose 1: number analyzed (Participants) | 365 | 119 | 121
  Any Fatigue, Dose 1 | 101 | 30 | 33
  Any Temperature (Axillary), Dose 1: number analyzed (Participants) | 365 | 119 | 121
  Any Temperature (Axillary), Dose 1 | 9 | 1 | 0
  Any Gastrointestinal symptoms, Dose 1: number analyzed (Participants) | 365 | 119 | 121
  Any Gastrointestinal symptoms, Dose 1 | 44 | 10 | 15
  Any Headache, Dose 1: number analyzed (Participants) | 365 | 119 | 121
  Any Headache, Dose 1 | 88 | 26 | 32
  Any Fatigue, Dose 2: number analyzed (Participants) | 361 | 0 | 118
  Any Fatigue, Dose 2 | 47 |  | 15
  Any Temperature (Axillary), Dose 2: number analyzed (Participants) | 361 | 0 | 118
  Any Temperature (Axillary), Dose 2 | 4 |  | 1
  Any Gastrointestinal symptoms, Dose 2: number analyzed (Participants) | 361 | 0 | 118
  Any Gastrointestinal symptoms, Dose 2 | 28 |  | 8
  Any Headache, Dose 2: number analyzed (Participants) | 361 | 0 | 118
  Any Headache, Dose 2 | 49 |  | 13
  Any Fatigue, Dose 3: number analyzed (Participants) | 359 | 0 | 116
  Any Fatigue, Dose 3 | 63 |  | 21
  Any Temperature (Axillary), Dose 3: number analyzed (Participants) | 359 | 0 | 116
  Any Temperature (Axillary), Dose 3 | 6 |  | 3
  Any Gastrointestinal symptoms, Dose 3: number analyzed (Participants) | 359 | 0 | 116
  Any Gastrointestinal symptoms, Dose 3 | 21 |  | 7
  Any Headache, Dose 3: number analyzed (Participants) | 359 | 0 | 116
  Any Headache, Dose 3 | 53 |  | 23
  Any Fatigue, Across doses: number analyzed (Participants) | 366 | 0 | 122
  Any Fatigue, Across doses | 149 |  | 48
  Any Temperature (Axillary), Across doses: number analyzed (Participants) | 366 | 0 | 122
  Any Temperature (Axillary), Across doses | 17 |  | 4
  Any Gastrointestinal symptoms, Across doses: number analyzed (Participants) | 366 | 0 | 122
  Any Gastrointestinal symptoms, Across doses | 72 |  | 23
  Any Headache, Across doses: number analyzed (Participants) | 366 | 0 | 122
  Any Headache, Across doses | 126 |  | 48

21. Secondary Outcome: Number of Subjects Reporting Any Unsolicited Adverse Events (AEs)
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: Up to 1 month after each vaccine dose
Population: The analysis was performed on the Total Vaccinated Cohort including all subjects with study vaccine administered.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Twinrix Group | Nimenrix Group | Twinrix Group
Number analyzed (Participants) | 367 | 122 | 122
Participants
  Post Dose 1 | 62 | 13 | 18
  Post Dose 2 | 26 | NA — Subjects in the Nimenrix Group only received 1 dose of vaccine. Hence, no results are available for Post Dose 2. | 7
  Post Dose 3 | 52 | NA — Subjects in the Nimenrix Group only received 1 dose of vaccine. Hence, no results are available for Post Dose 3. | 16

22. Secondary Outcome: Number of Subjects Reporting Any Specific AEs of New Onset of Chronic Illnesses
Description: Specific AEs of new onset of chronic illnesses include e.g. autoimmune disorders, asthma, type I diabetes and allergies.
Time Frame: During the entire study (up to Month 7)
Population: The analysis was performed on the Total Vaccinated Cohort including all subjects with study vaccine administered.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Twinrix Group | Nimenrix Group | Twinrix Group
Number analyzed (Participants) | 367 | 122 | 122
Participants | 5 | 0 | 2

23. Secondary Outcome: Number of Subjects Reporting Any Rash
Description: Rashes include e.g. hives, idiopathic thrombocytopenic purpura, petechiae.
Time Frame: During the entire study (up to Month 7)
Population: The analysis was performed on the Total Vaccinated Cohort including all subjects with study vaccine administered.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Twinrix Group | Nimenrix Group | Twinrix Group
Number analyzed (Participants) | 367 | 122 | 122
Participants | 5 | 0 | 1

24. Secondary Outcome: Number of Subjects Reporting Any Conditions Prompting Emergency Room Visits
Time Frame: During the entire study (up to Month 7)
Population: The analysis was performed on the Total Vaccinated Cohort including all subjects with study vaccine administered.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Twinrix Group | Nimenrix Group | Twinrix Group
Number analyzed (Participants) | 367 | 122 | 122
Participants | 1 | 0 | 0

25. Secondary Outcome: Number of Subjects Reporting Any Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: During the entire study (up to Month 7)
Population: The analysis was performed on the Total Vaccinated Cohort including all subjects with study vaccine administered.
Measure: Count of Participants; unit: Participants
Arm/Group | Nimenrix + Twinrix Group | Nimenrix Group | Twinrix Group
Number analyzed (Participants) | 367 | 122 | 122
Participants | 4 | 0 | 1

ADVERSE EVENTS:
Time Frame: Serious Adverse Events were reported throughout the entire study period (up to Month 7). Unsolicited Adverse Events were reported up to one month after each vaccine dose. Other Frequent (non-serious) Adverse Events were reported during a 4-day follow-up period after any vaccine dose.
Description: Other Frequent (non-serious) Adverse Events were reported only for those subjects who received the vaccination and completed their symptom sheet.
Arm/Group | Nimenrix + Twinrix Group | Nimenrix Group | Twinrix Group
All-Cause Mortality (participants affected / at risk) | 0/367 | 0/122 | 0/122
Serious Adverse Events (participants affected / at risk) | 4/367 | 0/122 | 1/122
Other Adverse Events (participants affected / at risk) | 312/367 | 82/122 | 100/122
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nimenrix + Twinrix Group (N=367) | Nimenrix Group (N=122) | Twinrix Group (N=122)
Brain contusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Drug toxicity (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Nimenrix + Twinrix Group (N=367) | Nimenrix Group (N=122) | Twinrix Group (N=122)
Pain at the injection site (General disorders) | 181 | 58 | 0/0 — Post-meningococcal vaccination
Swelling at the injection site (General disorders) | 62 | 18 | 0/0 — Post-meningococcal vaccination
Redness at the injection site (General disorders) | 75 | 19 | 0/0 — Post-meningococcal vaccination
Fatigue (General disorders) | 149 | 30 | 48
Gastrointestinal symptoms (General disorders) | 72 | 10 | 23
Headache (General disorders) | 126 | 26 | 48
Pain at the injection site (General disorders) | 228 | 0 | 73 — Post-Twinrix vaccination
Swelling at the injection site (General disorders) | 49 | 0 | 19 — Post-Twinrix vaccination
Redness at the injection site (General disorders) | 63 | 0 | 19 — Post-Twinrix vaccination

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.